CLINICAL TRIAL: NCT05995561
Title: Heidelberg Registry of Atrial Fibrillation
Brief Title: HERA FIb Registry for Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Mustafa Yildirim, Principle investigator, University Hospital Heidelberg
Other Study IDs: HERA FIb registry
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- atrial fibrillation: cases presenting with atrial fibrillation at the emegency department.
  Interventions: Other: no intervention is planned.

INTERVENTIONS:
Other: no intervention is planned. — no intervention is planned.

SUMMARY:
The single-center HERA AFIb registry was created to assess real-world prevalence, demographic characteristics and management of patients with atrial fibrillation (AF) in the era of novel oral anticoagulant regimes (NOAC) presenting in the emergency department (ED) of University of Heidelberg

DETAILED DESCRIPTION:
HERA AFIb is a single-center retrospective registry which enrolled consecutive cases presenting with atrial fibrillation at the emergency department of University Hospital of Heidelberg. Clinical parameters and characteristics for cases were assessed retrospectively. Follow-up was performed via review of medical reports, phone calls and postal queries. Outcome parameters included rates for all-cause mortality, non-hemorrhagic stroke, myocardial infarction and major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* documented atrial fibrillation
* availability of at least one hsTnT measurement

Exclusion Criteria:

* lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of approximately 13000 consecutive patients with atrial fibrillation presenting to the emergency department of the Heidelberg University Hospital.
Sampling Method: Probability Sample
Enrollment: 12297 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
all-cause mortality | 24 months
  all-cause mortality during follow-up

SECONDARY OUTCOMES:
ischaemic stroke | 24 months
  ischaemic stroke during follow-up
major bleeding | 24 months
  major bleeding during follow-up
myocardial infarction | 24 months
  myocardial infarction during follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salbach C, Yildirim M, Hund H, Muller-Hennessen M, Frey N, Katus HA, Giannitsis E, Milles BR. Effect of non-invasive rhythm control on outcomes in patients with first diagnosed atrial fibrillation presenting to an emergency department. BMC Emerg Med. 2025 Mar 3;25(1):35. doi: 10.1186/s12873-025-01194-z. PMID 40033211
- [Derived] Yildirim M, Milles BR, Hund H, Biener M, Muller-Hennessen M, Frey N, Katus HA, Giannitsis E, Salbach C. Outcomes and Disease Management in Patients With Atrial Fibrillation >/=80 Years: Data From a Consecutive 11-Year Real-World Registry. J Am Heart Assoc. 2025 Feb 18;14(4):e036832. doi: 10.1161/JAHA.124.036832. Epub 2025 Feb 8. PMID 39921512
- [Derived] Salbach C, Yildirim M, Hund H, Biener M, Muller-Hennessen M, Frey N, Katus HA, Giannitsis E, Milles BR. Design, Rationale and Initial Findings From HERA-FIB on 10 222 Patients With Atrial Fibrillation Presenting to an Emergency Department Over An 11-Year Period. J Am Heart Assoc. 2024 May 7;13(9):e033396. doi: 10.1161/JAHA.123.033396. Epub 2024 Apr 19. PMID 38639359